CLINICAL TRIAL: NCT00681980
Title: Study Of Valproic Acid To Treat TSP/HAM Patients In Sao Paulo, Brazil
Brief Title: Use Of Valproid Acid To Treat Tropical Spastic Paraparesis/HTLV-1-Associated Myelopathy (TSP/HAM)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Jorge Casseb, Professor, University of Sao Paulo
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 278
Record Dates: First submitted 2008-05-19; First posted 2008-05-21 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Paraparesis Spastic Tropical
Keywords: TSP/HAM, HTLV-1, treatment
MeSH Terms: conditions — Paraparesis, Tropical Spastic | interventions — Valproic Acid; Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A, 2, III (Experimental): Patients with side effects to corticosteroids
  Interventions: Drug: Valproic acid
- B (Experimental): patient with corticosteroids
  Interventions: Drug: costicosteroids
- 3 (Experimental): Valproic acid and corticosteroids
  Interventions: Drug: valproid acid plus corticosteroids

INTERVENTIONS:
Drug: Valproic acid — 15 mg/kg/day
  Arms: A, 2, III
Drug: costicosteroids — metypredsolone 1 g/day
  Arms: B
Drug: valproid acid plus corticosteroids — valporid acid 15 mg/kg/day plus corticosteroids 1 g/patient
  Arms: 3

SUMMARY:
Is the valproic acid efficacy to treat TSP/HAM

ELIGIBILITY:
Inclusion Criteria:

* HTLV-1; TSP/HAM fulfill criteria

Exclusion Criteria:

* Age <18 years

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-02; Primary Completion 2009-09 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Neurological sacles | 24 months

SECONDARY OUTCOMES:
Quality of life | 2009

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Tropical Medicine at Sao Paulo University, São Paulo, São Paulo, Brazil

REFERENCES:
- See also: Related Info — http://www.htlv.com.br